CLINICAL TRIAL: NCT01284907
Title: Vit D to Treat Asthma in Children: a Randomized, Double-blind, Placebo-controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Participants
Sponsor: United Arab Emirates University (Other)
Collaborators: Roma Paediatrics (Unknown)
Responsible Party: Dr Mariam Elremeli, Roma Paediatrics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMDHREC NO: 09/58
Record Dates: First submitted 2011-01-24; First posted 2011-01-27 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Asthma
Keywords: Asthma; Asthma therapy; Randomized controlled trial; children
MeSH Terms: conditions — Asthma | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vit D (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D3 (Cholecalciferol)
- Placebo drops (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Drops

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (Cholecalciferol) — Vit D3 ( Cholecalciferol) 1200 IU oral daily for 6 months
  Other Names: Cholecalciferol
  Arms: Vit D
Dietary Supplement: Placebo Drops
  Arms: Placebo drops

SUMMARY:
The purpose of this study is to determine whether vitamin D supplements can improve asthma control in children with moderate to severe asthma

DETAILED DESCRIPTION:
The proposed interventional study will clarify the role of vitamin D in preventing asthma exacerbations and in achieving better chronic asthma control in children with moderate to severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthmatics and they should fulfill at least two of the following three criteria:

  * A minimum of three clinic visits for acute asthma within 1 year
  * Two or more asthma-related hospital admissions within 1 year, or
  * Steroid dependency, as defined by either 6 months of oral or 1 year of inhaled corticosteroid use
* Age: 6-14 years old. The age group of 6 to 14 years old was chosen for two reasons:

  1. Diagnostic accuracy of asthma is better in this age group as non-specific wheezers less than 6 years of age could be excluded.
  2. Child should be able to use a peak flow meter and perform spirometry tests.
* A positive specific IgE or a positive skin prick test for at least one airborne allergen.

Exclusion Criteria:

* Children with mild intermittent and mild persistent asthma.
* Asthmatic children who are currently on immunotherapy or anti IgE.
* Asthmatic children with concomitant other medical problems.
* Children who are younger than 6 yrs or older than 14 yrs.
* Children with history of early life injury to airways like premature birth (< 36 weeks) or home use of oxygen.
* Children with vitamin D deficiency. Since these children may be randomized to the control group, they will be excluded for ethical reasons.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
A change from baseline in Peak expiratory flow rate | up to six months

SECONDARY OUTCOMES:
A change from baseline in lung function test | up to six months

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Elremeli, MD, Principal Investigator — Roma Paediatrics
Locations (2):
- United Arab Emirates (2):
  - Tawam Hospital, Al Ain City
  - Al Ain Hospital, Al Ain City